CLINICAL TRIAL: NCT07174245
Title: Pregnancy and Postpartum Continuous Glucose Monitoring in Gestational Diabetes
Brief Title: Pregnancy and Postpartum CGM in GDM
Status: Recruiting | Type: Observational
Sponsor: Icahn School of Medicine at Mount Sinai (Other)
Responsible Party: Principal Investigator, Grenye O'Malley, Associate Professor, Icahn School of Medicine at Mount Sinai
Other Study IDs: STUDY-25-00534
Record Dates: First submitted 2025-09-08; First posted 2025-09-15 (Actual); Last update posted 2025-09-15 (Actual); Status verified 2025-09

CONDITIONS: Gestational Diabetes
Keywords: gestational diabetes; continuous glucose monitor; glucose sensor; oral glucose tolerance test
MeSH Terms: conditions — Diabetes, Gestational

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (1):
- Participants with Gestational diabetes GDM: All participants who wear CGM and have their postpartum OGTT
  Interventions: Device: continuous glucose monitor

INTERVENTIONS:
Device: continuous glucose monitor — All participants who wear CGM
  Other Names: CGM

SUMMARY:
Gestational diabetes (GDM) is one of the most common complications of pregnancy, and up to one third of women with GDM will have abnormal blood sugars after their pregnancy. To screen for abnormal blood sugars, standard of care is a 4-12 week postpartum oral glucose tolerance test (OGTT). However only 17-60% of women actually have this test performed. This study is to assess continuous glucose monitor data from the third trimester and up to 14 days postpartum to find predictors of postpartum OGTT results.

DETAILED DESCRIPTION:
Those with GDM in current pregnancy using a Dexcom Continuous Glucose Monitoring (CGM) are eligible for enrollment. Participants use their CGM as usual during pregnancy and wear one sensor postpartum. They have their standard of care OGTT performed at around 6 weeks. They then complete a remote questionnaire after OGTT.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of gestational diabetes during current pregnancy
* age 18 or older
* prescribed Dexcom G7

Exclusion Criteria:

* Pregestational diabetes
* known skin adhesive allergy which inhibits ongoing use of CGM
* chronic oral steroid use.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Diagnosis of gestational diabetes during current pregnancy, age 18 or older, and prescribed Dexcom G7
Sampling Method: Non-Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2025-08-05 (Actual); Primary Completion 2026-08-05 (Estimated); Study Completion 2026-08-15 (Estimated)

PRIMARY OUTCOMES:
Sensitivity of postpartum TIR <96% | up to 12 weeks postpartum
  Sensitivity of postpartum time in range (TIR) <96% to predict dysglycemia on OGTT. Range 70-180 mg/dL.
  Sensitivity determined by true positives of TIR <96% and abnormal OGTT and false negatives would be TIR <96% with normal OGTT.

SECONDARY OUTCOMES:
Specificity of postpartum TIR <96% | up to 12 weeks postpartum
  Specificity of postpartum TIR <96% to predict dysglycemia on OGTT
  Specificity calculated by true negatives are TIR not <96% and normal OGTT and false positive are TIR <96% but normal OGTT results.
Experience survey questionnaire | up to 12 weeks postpartum
  6 items in non validated questionnaire to be administered remotely. first 5 questions rated on a 5 point likert scale. question 6 asks participant to choose preference between glucose sensor or oral glucose tolerance test.
  Each question evaluated on its own scored 1 (Strongly disagree) to 5 (Strongly Agree). The questions are not summed.

CONTACTS AND LOCATIONS:
Overall Officials: Grenye O'Malley, MD, Principal Investigator — Icahn School of Medicine at Mount Sinai
Locations (1):
- Icahn School of Medicine at Mount Sinai, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No
Identifying dates